CLINICAL TRIAL: NCT03831321
Title: The Effect of Preemptive Analgesia On The Comfort Of Patient and Doctor, in Cystoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taha Uçar (Other)
Responsible Party: Sponsor-Investigator, Taha Uçar, Resident Doctor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MedeniyetUro
Record Dates: First submitted 2019-01-01; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Bladder Cancer; Benign Prostate Hyperplasia; Hematuria; Pain; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Hyperplasia; Hematuria; Pain; Lower Urinary Tract Symptoms | interventions — Diclofenac; Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diclofenac group (Active Comparator): The group who are 50 mg Diclofenac Sodium and lubricant gel administered one hour before cystoscopy and local
  Interventions: Drug: Diclofenac Sodium; Device: Cystoscopy; Drug: Lubricant Gel
- Placebo (Placebo Comparator): The group who are not administered 50 mg Diclofenac Sodium before cystoscopy and administered lubricant gel just before local cystoscopy
  Interventions: Device: Cystoscopy; Drug: Lubricant Gel

INTERVENTIONS:
Drug: Diclofenac Sodium — 50 mg of diclofenac sodium will be administered to intervention group one hour before cystoscopy and lubricant gel with lidocaine will be administered to all patients just before cystoscopy.
  Arms: Diclofenac group
Device: Cystoscopy — Diagnostic cystoscopy
Drug: Lubricant Gel — To prevent patients from side effects of cystoscopy ( like urethral strictures and discomfort)

SUMMARY:
The study was designed as a prospective, randomized double-blind placebo controlled trial. According to power analysis in regards of previous studies in the literature with diclofenac sodium, using a total of 144 patients are needed for Power: 80% and Efficacy: 0.05. diclofenac (20 mg) and placebo drugs to be used in the study will be numbered 1 and 2 individually. Patient randomization was performed using random.org in 144 patients. On the day of cystoscopy, the patient randomized according to inclusion criteria will be given a medication package corresponding to the number given in randomization. It will not be known by the staff and cystoscopy will be performed by the physician who does not know which package is an effective drug.

Parameters:

1. Visual Pain Score during cystoscopy
2. Cystoscopy comfort - a questionnaire to be filled by the doctor

   1. Excellent
   2. Very good
   3. Good
   4. Bad
   5. Too bad
3. Cystoscopy: Is it efficient? Not efficient? - Will be answered by the doctor.

Post-Op:

1. 1st hour Visual Analog Pain Scale inquiry, dysuria, frequency
2. 24th Hour dysuria, Frequency,

A total of 144 patients, we plan to arrive at the end of 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Accepted to participate
* 18-70 years old
* Men

Exclusion Criteria:

1. Previous peptic ulcer
2. Gastro intestinal bleeding in advance
3. Renal failure
4. Liver failure
5. Patients who underwent cystoscopy for taking or inserting Double J stents 6 - Drug allergies

7- Patients under 18 8- Patients receiving antiaggregant and antiplatelet therapy 9- Patients who do not agree to participate in the study

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-04-22 (Estimated); Study Completion 2019-05-22 (Estimated)

PRIMARY OUTCOMES:
Assesment for operational pain | 1 minute
  All the patients will be assessed with Visual pain scale during cystoscopy procedure Scale is a well know pain assesment form which is ranged between 0 to 10 points and higher scores mean worse pain.

SECONDARY OUTCOMES:
Assesment of doctors comfort for the procedure(cystoscopy) | 1 minute
  It is subjective, It will made by a question which will be graded by the blind operator.
  The operator will choose one of the 5 answers. Scoring system will be range 1 to 5 and higher scores mean worse results.
Assesment of qualification of cystoscopy | 1 minute
  It is subjective. It will be made by a question which will be answered by blind operator.
  The operator will choose one of the answers which are "adequate or not adequate".

CONTACTS AND LOCATIONS:
Overall Officials: Asıf Yıldırım, Study Director — Medeniyet University
Locations (1):
- Medeniyet University, Istanbul, Outside U.S./Canada, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided